CLINICAL TRIAL: NCT02443909
Title: Comparison of Safety and Efficiency of 20w and 30w Holmium Laser Device in Management of 2-3 cm Diameter Kidney Stones With Retrograde Intrarenal Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, Nihat Karakoyunlu, MD, Diskapi Teaching and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 26.01.2015
Record Dates: First submitted 2015-04-28; First posted 2015-05-14 (Estimated); Last update posted 2015-05-14 (Estimated); Status verified 2015-05

CONDITIONS: Nephrolithiasis
Keywords: Holmium Laser; Kidney Stones; RIRS
MeSH Terms: conditions — Nephrolithiasis; Kidney Calculi

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- first group (Active Comparator): Patients undergoing Retrograde Intrarenal Surgery with 20w Holmium laser device who have 2-3 cm kidney stones
  Interventions: Procedure: Retrograde Intrarenal Surgery; Device: Holmium laser device
- second group (Active Comparator): Patients undergoing Retrograde Intrarenal Surgery with 30w Holmium laser device(working over 20w power) who have 2-3 cm kidney stones
  Interventions: Procedure: Retrograde Intrarenal Surgery; Device: Holmium laser device
- third group (Active Comparator): Patients undergoing Retrograde Intrarenal Surgery with 30w Holmium laser device(working under 20w power) who have 2-3 cm kidney ston
  Interventions: Procedure: Retrograde Intrarenal Surgery; Device: Holmium laser device

INTERVENTIONS:
Procedure: Retrograde Intrarenal Surgery — endoscopic stone treatment with flexible ureteroscopy and 20w holmium laser device
  Other Names: RIRS
  Arms: first group
Procedure: Retrograde Intrarenal Surgery — Retrograde Intrarenal Surgery with 30w Holmium laser device(working over 20w power)
  Other Names: RIRS
  Arms: second group
Procedure: Retrograde Intrarenal Surgery — Retrograde Intrarenal Surgery with 30w Holmium laser device(working under 20w power)
  Other Names: RIRS
  Arms: third group
Device: Holmium laser device

SUMMARY:
To compare safety and efficiency of 20w 30w holmium laser device in treatment of 2-3 cm diameter kidney stones with Retrograde Intrarenal Surgery (RIRS).

ELIGIBILITY:
Inclusion Criteria:

* patients who have 2-3 cm kidney stones
* patients who are between 18-90 years old

Exclusion Criteria:

* patients who have congenital urogenital abnormalities
* patients who have previous surgery history for urinary stones

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-12 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Safety (Complications according to clavien system) | 1 day
  Complications according to clavien system
Efficiency (visual analog score) | 1 Day
  visual analog score

SECONDARY OUTCOMES:
Efficiency (stone free rate) | 3 month
  stone free rate/

CONTACTS AND LOCATIONS:
Overall Officials: Nihat Karakoyunlu, MD, Principal Investigator — Ministry of Health, Turkey
Locations (1):
- S.B.Dıskapı Yıldırım Beyazıt Training and Research Hospital, Ankara, Turkey (Türkiye)

REFERENCES:
- [Result] Redondo C, Ramon de Fata F, Gimbernat H, Meilan E, Andres G, Angulo JC. Retrograde intrarenal surgery with holmium-YAG laser lithotripsy in the primary treatment of renal lithiasis. Actas Urol Esp. 2015 Jun;39(5):320-6. doi: 10.1016/j.acuro.2014.06.004. Epub 2014 Oct 25. English, Spanish. PMID 25443519